CLINICAL TRIAL: NCT06455254
Title: A Single-arm, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of Candonilimab（AK104） Combined With Regorafenib For the Third-line Treatment of MSS Colorectal Liver Metastasis
Brief Title: Cadonilimab Combined With Regorafenib as A Third-line Treatment in Patients With MSS CRLM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jin-hong Chen (Other)
Responsible Party: Sponsor-Investigator, Jin-hong Chen, Director, Clinical Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REGOCADO01
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: CRC
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Candonilimab (AK104) + Regorafenib
  Interventions: Drug: Candonilimab (AK104); Drug: Regorafenib

INTERVENTIONS:
Drug: Candonilimab (AK104) — Cadonilimab (AK104): 6mg/kg, i.v. q2w.
Drug: Regorafenib — Regorafenib: 80 mg p.o. qd for 3 weeks of every 4 week cycle (i.e. 3 weeks on, 1 week off).

SUMMARY:
This study is a single-arm, open-label, multicenter clinical study to evaluate the efficacy and safety of Candonilimab (AK104) combined with Regorafenib for the treatment of MSS colorectal liver metastasis. Candonilimab (AK104) is a humanized IgG1 bispecific antibody that targets PD-1 and CTLA-4.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter clinical study to evaluate the efficacy and safety of Candonilimab (AK104) combined with Regorafenib for the treatment of MSS colorectal liver metastasis. The purpose of the study is to observe and evaluate the efficacy and safety of Cadonilimab in combination with Regorafenib in patients with CRLM who had failed the previous second-line standard regimen, and to explore biomarkers related to efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old and < 75 years old;
* ECOG Performance status score 0 or 1;
* Histologically or cytologically confirmed adenocarcinoma of colon or rectum, with liver metastases, with or without extrahepatic metastases;
* At least one measurable lesion as defined by RECIST version 1.1;
* Progressed or be intolerant to prior systemic therapy including fluoropyrimidines, irinotecan, oxaliplatin, bevacizumab and/or cetuximab/panitumumab (if RAS/RAF-wild-type);
* Known RAS and BRAF status;
* Only patients with mismatch repair-proficient (pMMR)/microsatellite stable (MSS) status;
* Adequate bone-marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 7 days of starting to study treatment:

Liver and renal function: Total bilirubin ≤ 1.5× ULNl; aspartate transaminase (AST), alanine transaminase (ALT) ≤ 5× ULN; Serum creatinine ≤ 1.5× ULN; Bone-marrow function: Neutrophil count ≥ 1.5×10^9/L, Hemoglobin (Hb) ≥ 9.0 g/dL, Platelet count ≥ 100×10^9/L; International normalised ratio (INR) and partial thromboplastin time (PTT) ≤1.5 × ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of an underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care；

* Patients of childbearing potential must be willing to use highly effective contraception for the duration of the study and for ≥120 days after the last dose of cadonilimab; female patients with a negative urine or serum pregnancy test result within ≤3 days prior to the first dose of the drug;
* Able to understand and voluntarily sign written informed consent;
* No history of allergy to regorafenib, cadonilimab and its components.

Exclusion Criteria:

* Women who are pregnant or breastfeeding;
* Patients who have previously been treated with third-line regimens such as regorafenib, fruquintinib, trifluridine tipiracil, or other immune checkpoint inhibitors, including anti-PD-1, anti-PD-L1, anti-CTLA-4, or any cellular immunotherapy;
* Active autoimmune disease requiring systemic therapy within the past 2 years (e.g., treatment with disease-modifying drugs, corticosteroids, immunosuppressants), replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid therapy for adrenal or pituitary insufficiency) is not considered a systemic treatment;
* Active or prior history of definite inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea);
* Patients who have received intervention, ablation or radiotherapy within the previous 3 months for the target lesion;
* Patients with an expected survival time of less than 3 months;
* Study participants with other malignant tumors within 3 years prior to enrollment, excluding cured local tumors (such as basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, etc.);
* Patients with severe psychological or psychiatric abnormalities;
* No history of severe arrhythmia, heart failure, severe ventilatory dysfunction and severe lung infection, no acute and chronic renal failure;
* Concurrent enrollment in another clinical study, unless it is an observational, non-interventional clinical study or a follow-up period of an interventional study;
* Any other clinically significant disease or condition that, in the opinion of the investigator, may affect adherence to the protocol, or the signing of the Informed Consent Form (ICF) by the subject, or make participation in this clinical trial inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  ORR, determined using RECIST v1.1, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 6 months
  DCR, determined using RECIST v1.1, defined as the percentage of subjects whose best response was not PD (= total number of CR + PR + SD; CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating)
Duration of response (DoR) | 6 months
  DoR, determined using RECIST v1.1, defined as the time from the first judgment of CR or PR to the discovery of PD after treatment.
Progression-free Survival (PFS) | 6 months
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.
Overall survival (OS) | 2 years
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Adverse event incidence rate (AE rate) | 6 months
  Safety variables will be summarized using descriptive statistics based on adverse events collection.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Huashan Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Data are available from the corresponding author on reasonable request.
Time Frame: Up to 1 year after the end of the study.
Access Criteria: Applicants contact researchers by email to obtain data.

REFERENCES:
- [Background] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Background] Siegel RL, Wagle NS, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2023. CA Cancer J Clin. 2023 May-Jun;73(3):233-254. doi: 10.3322/caac.21772. Epub 2023 Mar 1. PMID 36856579
- [Background] Li J, Qin S, Xu R, Yau TC, Ma B, Pan H, Xu J, Bai Y, Chi Y, Wang L, Yeh KH, Bi F, Cheng Y, Le AT, Lin JK, Liu T, Ma D, Kappeler C, Kalmus J, Kim TW; CONCUR Investigators. Regorafenib plus best supportive care versus placebo plus best supportive care in Asian patients with previously treated metastatic colorectal cancer (CONCUR): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):619-29. doi: 10.1016/S1470-2045(15)70156-7. Epub 2015 May 13. PMID 25981818
- [Background] Li J, Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Fan S, Hua Y, Su W. Effect of Fruquintinib vs Placebo on Overall Survival in Patients With Previously Treated Metastatic Colorectal Cancer: The FRESCO Randomized Clinical Trial. JAMA. 2018 Jun 26;319(24):2486-2496. doi: 10.1001/jama.2018.7855. PMID 29946728
- [Background] Dasari A, Lonardi S, Garcia-Carbonero R, Elez E, Yoshino T, Sobrero A, Yao J, Garcia-Alfonso P, Kocsis J, Cubillo Gracian A, Sartore-Bianchi A, Satoh T, Randrian V, Tomasek J, Chong G, Paulson AS, Masuishi T, Jones J, Csoszi T, Cremolini C, Ghiringhelli F, Shergill A, Hochster HS, Krauss J, Bassam A, Ducreux M, Elme A, Faugeras L, Kasper S, Van Cutsem E, Arnold D, Nanda S, Yang Z, Schelman WR, Kania M, Tabernero J, Eng C; FRESCO-2 Study Investigators. Fruquintinib versus placebo in patients with refractory metastatic colorectal cancer (FRESCO-2): an international, multicentre, randomised, double-blind, phase 3 study. Lancet. 2023 Jul 1;402(10395):41-53. doi: 10.1016/S0140-6736(23)00772-9. Epub 2023 Jun 15. PMID 37331369
- [Background] Fukuoka S, Hara H, Takahashi N, Kojima T, Kawazoe A, Asayama M, Yoshii T, Kotani D, Tamura H, Mikamoto Y, Hirano N, Wakabayashi M, Nomura S, Sato A, Kuwata T, Togashi Y, Nishikawa H, Shitara K. Regorafenib Plus Nivolumab in Patients With Advanced Gastric or Colorectal Cancer: An Open-Label, Dose-Escalation, and Dose-Expansion Phase Ib Trial (REGONIVO, EPOC1603). J Clin Oncol. 2020 Jun 20;38(18):2053-2061. doi: 10.1200/JCO.19.03296. Epub 2020 Apr 28. PMID 32343640
- [Background] Cousin S, Cantarel C, Guegan JP, Gomez-Roca C, Metges JP, Adenis A, Pernot S, Bellera C, Kind M, Auzanneau C, Le Loarer F, Soubeyran I, Bessede A, Italiano A. Regorafenib-Avelumab Combination in Patients with Microsatellite Stable Colorectal Cancer (REGOMUNE): A Single-arm, Open-label, Phase II Trial. Clin Cancer Res. 2021 Apr 15;27(8):2139-2147. doi: 10.1158/1078-0432.CCR-20-3416. Epub 2021 Jan 25. PMID 33495314
- [Background] Guo Y, Zhang W, Ying J, Zhang Y, Pan Y, Qiu W, Fan Q, Xu Q, Ma Y, Wang G, Guo J, Su W, Fan S, Tan P, Wang Y, Luo Y, Zhou H, Li J. Phase 1b/2 trial of fruquintinib plus sintilimab in treating advanced solid tumours: The dose-escalation and metastatic colorectal cancer cohort in the dose-expansion phases. Eur J Cancer. 2023 Mar;181:26-37. doi: 10.1016/j.ejca.2022.12.004. Epub 2022 Dec 13. PMID 36628898
- [Background] Frentzas S, Gan HK, Cosman R, Coward J, Tran B, Millward M, Zhou Y, Wang W, Xia D, Wang ZM, Li B, Xia M, Desai J. A phase 1a/1b first-in-human study (COMPASSION-01) evaluating cadonilimab in patients with advanced solid tumors. Cell Rep Med. 2023 Nov 21;4(11):101242. doi: 10.1016/j.xcrm.2023.101242. Epub 2023 Oct 17. PMID 37852261
- [Background] Gao X, Xu N, Li Z, Shen L, Ji K, Zheng Z, Liu D, Lou H, Bai L, Liu T, Li Y, Li Y, Fan Q, Feng M, Zhong H, Huang Y, Lou G, Wang J, Lin X, Chen Y, An R, Li C, Zhou Q, Huang X, Guo Z, Wang S, Li G, Fei J, Zhu L, Zhu H, Li X, Li F, Liao S, Min Q, Tang L, Shan F, Gong J, Gao Y, Zhou J, Lu Z, Li X, Li J, Ren H, Liu X, Yang H, Li W, Song W, Wang ZM, Li B, Xia M, Wu X, Ji J. Safety and antitumour activity of cadonilimab, an anti-PD-1/CTLA-4 bispecific antibody, for patients with advanced solid tumours (COMPASSION-03): a multicentre, open-label, phase 1b/2 trial. Lancet Oncol. 2023 Oct;24(10):1134-1146. doi: 10.1016/S1470-2045(23)00411-4. PMID 37797632